CLINICAL TRIAL: NCT03848819
Title: Effect of the VitaBreath Device on Chest Wall Dynamic Hyperinflation and Respiratory Muscle Activation During Recovery From Exercise in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Portable NIV on Operational Chest Wall Volumes in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: North Tyneside General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 259201
Record Dates: First submitted 2019-02-13; First posted 2019-02-21 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2019-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Dynamic Hyperinflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is a randomised crossover trial. Patients will perform two identical exercise tests and the intervention (VitaBreath) will be compared to control condition (pursed-lip breathing) in the same patients.The order of testing will be determined by simple randomisation (sealedenvelope.com).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control pursed lip breathing (Other): Patients will undergo one intermittent exercise protocols on a cycle ergometer. The exercise protocol will consist of repeated 2-min exercise bouts, separated by 2-min recovery periods in between work bouts. During the 1st min of each recovery period patients will breathe adopting the pursed lip breathing technique. During the 2nd min of each recovery period patients will breathe normally. Patients will also score the intensity of their perceived dyspnoea using the Borg 1-10 scale. Cardiac output and stroke volume will be measured non-invasively using a cardio-impedance method (physio-flow) throughout the exercise and recovery periods. Respiratory muscle activation (EMG) and local respiratory muscle oxygen tissue oxygenation (NIRS) will be continuously recorded non-invasively using optodes placed on the skin throughout the exercise and recovery periods. In addition, arterial oxygen saturation will be recorded throughout the exercise and recovery periods using a pulse oximeter.
  Interventions: Device: VitaBreath device
- pNIV (Experimental): Patients will undergo one intermittent exercise protocols on a cycle ergometer. The exercise protocol will consist of repeated 2-min exercise bouts, separated by 2-min recovery periods in between work bouts. During the 1st min of each recovery period patients will breathe via the VitaBreath device. During the 2nd min of each recovery period patients will breathe normally. Patients will also score the intensity of their perceived dyspnoea using the Borg 1-10 scale. Cardiac output and stroke volume will be measured non-invasively using a cardio-impedance method (physio-flow) throughout the exercise and recovery periods. Respiratory muscle activation (EMG) and local respiratory muscle oxygen tissue oxygenation (NIRS) will be continuously recorded non-invasively using optodes placed on the skin throughout the exercise and recovery periods. In addition, arterial oxygen saturation will be recorded throughout the exercise and recovery periods using a pulse oximeter.
  Interventions: Device: VitaBreath device

INTERVENTIONS:
Device: VitaBreath device — The VitaBreath (Philips, Respironics) is a portable, handheld, battery powered, non-invasive ventilation device, that has been shown by our group to reduce activity-related shortness of breath in patients with COPD. It delivers 18 cmH2O inspiratory and 8 cmH2O expiratory pressures, but can only be used during recovery periods. In our study patients will perform consecutive bouts of exercise alternated by two minute of recovery in order to allow the use of the VitaBreath device during the first minute of each recovery period.

SUMMARY:
The VitaBreath (Philips, Respironics) is a portable, handheld, battery powered, non-invasive ventilation device, that has been shown to reduce activity-related shortness of breath in patients with COPD. The VitaBreath device delivers 18 cmH2O inspiratory and 8 cmH2O expiratory pressures, but can only be used during recovery periods.

A previous study (REC: 17/NE/0085) showed that use of the VitaBreath device during the recovery periods interspersing successive exercise bouts enhances exercise tolerance and reduces breathlessness compared to pursed lip breathing in patients with COPD. This was attributed to faster recovery from exercise-induced dynamic hyperinflation, assessed by volitional inspiratory capacity manoeuvres using a spirometer. However, inspiratory capacity manoeuvres are effort dependent, thus limiting the number of repetitions the patient can perform during exercise. In addition, investigation of the direct effect of the application of the VitaBreath device on dynamic hyperinflation was not possible due to the need to employ a spirometer for assessing inspiratory capacity. Optoelectronic plethysmography (OEP) allows continuous non-invasive assessment of end-inspiratory and end-expiratory volumes of the thoracoabdominal wall and its compartments, thereby facilitating assessment of dynamic hyperinflation on a breath-by-breath basis without the necessity to breathe via a spirometer. Unfortunately, OEP technology was not available at the time of our previous study.

The investigators will use OEP to provide accurate breath-by-breath volume measurements during exercise and recovery to evaluate whether the VitaBreath device reduces total and compartmental thoracoabdominal wall volumes compared to the pursed lip breathing technique.

Furthermore, the investigators will investigate the effect of use of the VitaBreath device on respiratory muscle activation and respiratory muscle oxygenation using OEP technology in conjunction with electromyography (EMG) and near inferred spectroscopy (NIRS), respectively to appreciate how the application of the VitaBreath device impacts on the operation and energy demands of the respiratory muscles as compared to control pursed lip breathing.

The investigators hypothesised that the use of the VitaBreath device during the recovery periods interspersing successive exercise bouts will reduce the magnitude of dynamic hyperinflation in a greater extent compared to the pursed lip breathing technique.

DETAILED DESCRIPTION:
Study Design:

This is a randomised crossover trial. Patients will perform two identical exercise tests and the intervention (VitaBreath) will be compared to control condition (pursed-lip breathing) in the same patients. The order of testing will be determined by simple randomisation (sealedenvelope.com).

The purpose of this study is to investigate the effect of the VitaBreath device on inspiratory and expiratory thoracoabdominal wall volumes during exercise in patients with COPD. Use of the VitaBreath device will be compared to normal breathing (pursed lip breathing technique). Patients will primarily be recruited from those who participated in our previous study (REC reference: 17/NE/0085 - IRAS project ID: 221120) at North Tyneside General Hospital and will undergo two exercise tests on a cycle ergometer on the same day using both the VitaBreath device and the pursed-lip breathing technique during recovery from exercise.

Study interventions:

The study will include two visits. During the first visit patients will undergo a clinical assessment, including history, physical examination, ECG and full lung function assessment including spirometry, to ensure that patients are stable. During the second visit patients will perform two intermittent exercise tests lasting 20 minutes each and consisting of 2-min work bouts at 80% of peak work rate (WR peak) as determined in the previous study (REC reference: 17/NE/0085 - IRAS project ID: 221120) with 2-min recovery periods in between work bouts, using either the VitaBreath device or the pursed lip breathing technique during recovery periods. Patients will be given written information explaining the procedure and will provide written informed consent.

Assessment Procedures

Visit 1

Baseline assessment

During the first visit patients will undergo the following baseline assessment: a) medical history and physical examination, b) spirometry and c) resting ECG to assess the resting heart function.

Visit 2

Preparation of the patients

Upon arrival to the laboratory, and prior to any intervention, adhesive skin markers for Opto-Electronic Plethysmography (OEP) recordings (to assess thoracoabdominal wall dynamic hyperinflation), and set of adhesive optodes for portable cardio-impedance recordings (to assess cardiac output), muscle surface electromyography (to assess muscle recruitment patterns) and near inferred spectroscopy (to assess respiratory muscle oxygen requirement) will be attached on the skin. All procedures will be explained in detail prior each trial.

Operational chest wall volumes

At baseline, patients will be instructed after 3-4 regular tidal breaths to make two maximal inspiratory capacity (IC) efforts from End Expiratory Chest Wall (EECW) Volume to Total Chest Wall Capacity (TLCCW) in order to assess chest wall volume at TLC (TLCCW) and Inspiratory Reserve Chest wall Volume (IRVcw) at rest. During exercise and recovery, chest wall kinematics will be measured by OEP as follows: the movement of 89 retro-reflective markers placed front and back over the chest wall from clavicles to pubis will be recorded. Each marker will be tracked by eight video cameras (Smart System BTS, Milan, Italy), four in front of the subject and four behind. Subjects will be grasp handles positioned at the mid sternum level which will lift the arms away from the rib cage so that lateral markers can be visualised. Dedicated software reconstructs the three-dimensional coordinates of the markers in real time by stereophotogrametry and calculates total and compartmental chest wall volume and volume variations using Gauss's theorem. The chest wall is modelled as being composed of two compartments-the rib cage and the abdomen. Vcw is the sum of the rib cage volume (Vrc) and abdominal volume (Vab).

Non-Invasive assessment of respiratory muscle oxygenation

In addition to operational chest wall volumes investigators are going to assess intercostal and abdominal local muscle oxygenation using Near-Infrared Spectroscopy (NIRS). Two NIRS optodes, which will be connected to a NIRO 200 spectrophotometer (Hamamatsu Photonics, Hamamatsu, Japan), will be placed on the skin over the left seventh intercostal space at the midaxillary line and over the upper rectus abdominis respectively, and will be secured using adhesive tape. The left intercostal space will be used to avoid potential blood flow contributions from the liver on the right side of the body.

Respiratory muscle electromyography

Electromyography (EMG) will be used in order assess respiratory muscle activation. Skin will be cleaned and surface electrodes (Delsys Trigno, Delsys, Boston, MA, USA) will be placed as follows: on the surface over the right seventh intercostal space (EMGic), 2 cm lateral to the umbilicus, over the muscle mass of rectus abdominis (EMGra), over the sternocleidomastoid muscle (EMGster), and on the scalene muscle (EMGsca). EMG data will be recorded at 2000Hz and will be filtered at 25-500 Hz during each trial (Spike 2, Cambridge Electronic Design, Cambridge, UK).

Exercise protocol

Patients will undergo two intermittent exercise protocols on a cycle ergometer. The exercise protocol will consist of repeated 2-min exercise bouts, separated by 2-min recovery periods in between work bouts in order to allow application of the VitaBreath device. During the 1st min of each recovery period patients will breathe either via the VitaBreath device or adopting the pursed lip breathing technique. During the 2nd min of each recovery period patients will breathe normally. Patients will also score the intensity of their perceived dyspnoea using the Borg 1-10 scale. Cardiac output and stroke volume will be measured non-invasively using a cardio-impedance method (physio-flow) throughout the exercise and recovery periods. Respiratory muscle activation (EMG) and local respiratory muscle oxygen tissue oxygenation (NIRS) will be continuously recorded non-invasively using optodes placed on the skin throughout the exercise and recovery periods. In addition, arterial oxygen saturation will be recorded throughout the exercise and recovery periods using a pulse oximeter.

Sample size estimation

Estimation of sample size within each breathing modality is based on the results of a study comparing use of the VitaBreath device to pursed lip breathing (PLB). Using the mean difference in the recovery of inspiratory capacity compared to the end of exercise (130 ml) between the VitaBreath device and PLB, the SD (110 ml), an alpha significance level of 0.05 (2-sided) and 80% power, a minimum total sample size of 11 patients is calculated to be sufficient to detect significant differences in the magnitude of change in thoracoabdominal wall dynamic hyperinflation between the VitaBreath device and PLB trials. 12 patients will be recruited in order to perform the trials in a balanced ordering sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 40 years or older.
2. Current or previous smoking history: 10 or more pack years.
3. Spirometry confirmed stable COPD (GOLD stages II-IV) under optimal medical therapy.
4. Exhibit substantial exercise-induced dynamic hyperinflation (ΔIC baseline > 0,150 L)

Exclusion Criteria:

1. Orthopaedic, neurological or other concomitant diseases that significantly impair normal biomechanical movement patterns, as judged by the investigator.
2. Moderate or severe COPD exacerbation within 6 weeks.
3. Unstable cardiac arrhythmia.
4. Unstable ischaemic heart disease, including myocardial infarction within 6 weeks.
5. Moderate or severe aortic stenosis or hypertrophic obstructive cardiomyopathy.
6. Uncontrolled hypertension.
7. Uncontrolled hypotension (SBP<85mmHg).
8. Uncontrolled diabetes.
9. Intolerance of the VitaBreath device.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
The magnitude of change in thoracoabdominal wall dynamic hyperinflation. | The intervention will be performed in one visit. During the visit patients will perform 2 trials lasting for 20 minutes each. The outcome 1 will be assessed at rest, at the 20th minute of cycling and 5 minutes post cycling at each trial.
  Change from baseline in litres of thoracoabdominal wall volume at end of exercise and recovery from exercise from resting breathing.

SECONDARY OUTCOMES:
Compartmental thoracoabdominal wall volumes (rib cage and abdominal volumes) assessed by OEP. | The intervention will be performed in one visit. During the visit patients will perform 2 trials lasting for 20 minutes each. The outcome 2 will be assessed at rest, at the 20th minute of cycling and 5 minutes post cycling at each trial.
  Change from baseline in litres of compartmental thoracoabdominal wall volume at end of exercise and recovery from exercise from resting breathing.
Electromyographic activation (expressed as fractions of peak activation and in absolute terms in mV) assessed by surface electromyography | The intervention will be performed in one visit. During the visit patients will perform 2 trials lasting for 20 minutes each. The outcome 3 will be assessed at rest, at the 20th minute of cycling and 5 minutes post cycling at each trial.
  Change from baseline in integrated EMG signal from respiratory muscles at end of exercise and recovery from exercise from resting breathing.
Respiratory muscle oxygenation requirements recorded from the intercostal and abdominal muscles by near infrared spectroscopy including measurements of: total haemoglobin (TOI), oxygenated haemoglobin (HbO2) and deoxygenated haemoglobin (HHb). | The intervention will be performed in one visit. During the visit patients will perform 2 trials lasting for 20 minutes each. The outcome 4 will be assessed at rest, at the 20th minute of cycling and 5 minutes post cycling at each trial.
  Change from baseline in fractional oxygen saturation of the respiratory muscles at end of exercise and recovery from exercise from resting breathing.
Cardiac output responses assessed non-invasively by cardio impedance technology | The intervention will be performed in one visit. During the visit patients will perform 2 trials lasting for 20 minutes each. The outcome 5 will be assessed at rest, at the 20th minute of cycling and 5 minutes post cycling at each trial.
  Change from baseline in cardiac output at end of exercise and recovery from exercise from resting breathing.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Donnell DE, Revill SM, Webb KA. Dynamic hyperinflation and exercise intolerance in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Sep 1;164(5):770-7. doi: 10.1164/ajrccm.164.5.2012122. PMID 11549531
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Vogiatzis I, Zakynthinos S. Factors limiting exercise tolerance in chronic lung diseases. Compr Physiol. 2012 Jul;2(3):1779-817. doi: 10.1002/cphy.c110015. PMID 23723024
- [Background] Beauchamp MK, Nonoyama M, Goldstein RS, Hill K, Dolmage TE, Mathur S, Brooks D. Interval versus continuous training in individuals with chronic obstructive pulmonary disease--a systematic review. Thorax. 2010 Feb;65(2):157-64. doi: 10.1136/thx.2009.123000. Epub 2009 Dec 8. PMID 19996334
- [Background] Morris NR, Walsh J, Adams L, Alision J. Exercise training in COPD: What is it about intensity? Respirology. 2016 Oct;21(7):1185-92. doi: 10.1111/resp.12864. PMID 27623321
- [Background] Puente-Maestu L, Palange P, Casaburi R, Laveneziana P, Maltais F, Neder JA, O'Donnell DE, Onorati P, Porszasz J, Rabinovich R, Rossiter HB, Singh S, Troosters T, Ward S. Use of exercise testing in the evaluation of interventional efficacy: an official ERS statement. Eur Respir J. 2016 Feb;47(2):429-60. doi: 10.1183/13993003.00745-2015. Epub 2016 Jan 21. PMID 26797036
- [Background] Sabapathy S, Kingsley RA, Schneider DA, Adams L, Morris NR. Continuous and intermittent exercise responses in individuals with chronic obstructive pulmonary disease. Thorax. 2004 Dec;59(12):1026-31. doi: 10.1136/thx.2004.026617. PMID 15563700
- [Background] O'Donnell DE, D'Arsigny C, Webb KA. Effects of hyperoxia on ventilatory limitation during exercise in advanced chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Mar;163(4):892-8. doi: 10.1164/ajrccm.163.4.2007026. PMID 11282762
- [Background] Palange P. Lighter than air: heliox breathing improves exercise tolerance in COPD. Eur Respir Rev. 2010 Mar;19(115):1-3. doi: 10.1183/09059180.00000210. No abstract available. PMID 20956159
- [Background] Ambrosino N, Cigni P. Non invasive ventilation as an additional tool for exercise training. Multidiscip Respir Med. 2015 Apr 9;10(1):14. doi: 10.1186/s40248-015-0008-1. eCollection 2015. PMID 25874110
- [Background] Vogiatzis I, Chynkiamis N, Armstrong M, Lane ND, Hartley T, Gray WK, Bourke SC. Intermittent Use of Portable NIV Increases Exercise Tolerance in COPD: A Randomised, Cross-Over Trial. J Clin Med. 2019 Jan 15;8(1):94. doi: 10.3390/jcm8010094. PMID 30650617
- [Background] Vogiatzis I, Georgiadou O, Golemati S, Aliverti A, Kosmas E, Kastanakis E, Geladas N, Koutsoukou A, Nanas S, Zakynthinos S, Roussos C. Patterns of dynamic hyperinflation during exercise and recovery in patients with severe chronic obstructive pulmonary disease. Thorax. 2005 Sep;60(9):723-9. doi: 10.1136/thx.2004.039115. Epub 2005 Jun 17. PMID 15964912
- See also: Philips white paper — http://usermanual.wiki/Philips/vitabreathwhitepapera4final.3771554293.pdf